CLINICAL TRIAL: NCT01410409
Title: Structured Treatment of Osteoarthritis of the Knee With or Without Total Knee Replacement. A Randomized Controlled Trial of Pain, Physical Function and Quality of Life With 12months Follow-up
Brief Title: Structured Treatment of Osteoarthritis of the Knee With or Without Total Knee Replacement
Acronym: MEDIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Collaborators: The Danish Rheumatism Association (Other); Obel Family Foundation (Unknown); Spar Nord Foundation (Unknown); The Bevica Foundation (Unknown); Aalborg University (Other); Association of Danish Physiotherapists (Other); Formthotics (Unknown); Medical Specialist Heinrich Kopp's Grant (Unknown); Danish Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N-20110024
Record Dates: First submitted 2011-08-02; First posted 2011-08-05 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis, Knee; Treatment Outcome; Time Factors; Arthroplasty, Replacement; Rehabilitation; Combined Modality Therapy; Middle Aged; Aged; Aged, 80 and over; Male; Female; Humans; Analysis of Variance
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Acetaminophen; Pantoprazole; Nutrition Assessment; Patient Education as Topic; Arthroplasty, Replacement, Knee; Foot Orthoses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MEDIC (Active Comparator): Medicine, Exercise, Diet, Insole and Cognitive/patient education (MEDIC) for three months.
  Interventions: Other: Neuromuscular training (NEMEX-TJR); Drug: Paracetamol; Drug: Burana; Drug: Pantoprazol; Behavioral: Dietary counseling; Behavioral: Patient education; Other: Insoles
- MEDIC + TKR (Active Comparator): Medicine, Exercise, Diet, Insole and Cognitive/patient education (MEDIC) for three months after a total knee replacement.
  Interventions: Other: Neuromuscular training (NEMEX-TJR); Drug: Paracetamol; Drug: Burana; Drug: Pantoprazol; Behavioral: Dietary counseling; Behavioral: Patient education; Procedure: TKR; Other: Insoles
- Observational Cohort (Active Comparator): If the patient can be included, but doesn't want to participate in the randomization, the patient is offered to enter into a prospective observational cohort with the same endpoints and the same follow-up as in the randomized study. The participant can then, in consultation with his/her physician, choose whether they would like MEDIC-treatment or TKR in combination with MEDIC-treatment.
  Interventions: Other: Neuromuscular training (NEMEX-TJR); Drug: Paracetamol; Drug: Burana; Drug: Pantoprazol; Behavioral: Dietary counseling; Behavioral: Patient education; Procedure: TKR; Other: Insoles

INTERVENTIONS:
Other: Neuromuscular training (NEMEX-TJR) — 60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Other Names: no other names
Drug: Paracetamol — 1 g x 4/day
  Other Names: no other names
Drug: Burana — 400 mg x 3/day for three weeks
  Other Names: NSAIDs are chosen in collaboration with the participant.
Drug: Pantoprazol — 20mg x 1/day for three weeks
  Other Names: no other names
Behavioral: Dietary counseling — For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet and plans the number of visits according to the individual participant needs.
  Other Names: no other names
Behavioral: Patient education — The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA. This aspect of the intervention is based on principles from The Chronic Disease Self-Management Program, "Lær at leve med kronisk sygdom (Learn to live with chronic illness)" by The National Board of Health, Denmark and "Artrosskolan Spenshult" in Sweden.
  Other Names: no other names
Procedure: TKR — Surgical treatment with insertion of total knee replacement following standard procedures.
  Other Names: Total Knee Replacement; Knee arthroplasty
  Arms: MEDIC + TKR; Observational Cohort
Other: Insoles — The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
  The participants will be advised to use the insoles in all shoes.
  Other Names: no other names

SUMMARY:
The purpose of this study is to test whether surgical insertion of total knee replacement provides further improvement in quality of life, pain and function in addition to an algorithm for systematic non-surgical treatment consisting of corrective insoles, neuromuscular training, weight loss, patient education and pharmacological treatment with paracetamol, NSAIDs and Pantoprazol in patients with knee OA, collectively called the MEDIC-treatment(Medicine Exercise Diet Insoles Cognitive).

The H1-hypothesis is that surgery with insertion of TKR in addition to the MEDIC-treatment results in a greater increase in quality of life and functional capacity and greater reduction in pain than the MEDIC- treatment alone at the primary endpoint, which is follow-up 12months after the start of the treatment.

See statistical analysis plan available under "Links" for further description of the study.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the degenerative joint disease that most often requires treatment and at the same time the one associated with the greatest social costs. In addition, the disease has many personal costs and is greatly contributing to reduced functionality and autonomy of older adults.

It is recommended both nationally and internationally that the treatment of knee OA should include multiple treatment modalities. Clinical guidelines recommend that exercise, weight loss and patient education is the first step in treatment and that insoles and pharmacological treatment can be included as a supplement. If this non-surgical treatment is ineffective surgical treatment, especially surgery with insertion of total knee replacement (TKR), may be indicated. There are effects of both non-surgical treatment and TKR, but no studies exist, which examine the effect of surgery with insertion of TKR in addition to the recommended non-surgical treatment of knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Knee-OA detected by x-ray (Kellgren & Lawrence grade 2 or greater)
* Considered a candidate for TKR by the orthopedic surgeon.
* The participant is > 18 years of age.
* The participant can provide relevant and adequate, informed consent.

Exclusion Criteria:

* Bilateral simultaneous TKR
* Revision of prior TKR, unicompartmental knee arthroplasty or high tibial osteotomy
* Rheumatoid arthritis
* Mean VAS > 60mm on a 0-100mm scale
* Investigator considers that the mental condition of the participant does not allow participation.
* The participant must not be pregnant or plan pregnancy during the study.
* Inability to comply with the protocol;.
* Inadequacy in written and spoken Danish.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Søren T Skou, PhD-student, Principal Investigator — Orthopaedic Research Unit, Aalborg University Hospital, Denmark; Ewa M Roos, PhD, Study Chair — Institute of Sports Science and Clinical Biomechanics, University of Southern Denmark, Denmark; Lars Arendt-Nielsen, Dr.Sci.Med., Study Chair — Center for Sensory-Motor Interaction (SMI), Department of Health Sciences and Technology, Aalborg University; Mogens B Laursen, PhD, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Sten Rasmussen, MD, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Michael S Rathleff, PhD-student, Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark; Ole H Simonsen, Dr.Med., Study Chair — Orthopaedic Surgery Research Unit, Aalborg University Hospital, Denmark
Locations (3):
- Denmark (3):
  - Department of Occupational and Physiotherapy, Aalborg University Hospital, Aalborg
  - Farsoe Hospital, Farsø
  - Vendsyssel Hospital, Frederikshavn, Frederikshavn

REFERENCES:
- [Background] Peat G, McCarney R, Croft P. Knee pain and osteoarthritis in older adults: a review of community burden and current use of primary health care. Ann Rheum Dis. 2001 Feb;60(2):91-7. doi: 10.1136/ard.60.2.91. PMID 11156538
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Jordan KM, Arden NK, Doherty M, Bannwarth B, Bijlsma JW, Dieppe P, Gunther K, Hauselmann H, Herrero-Beaumont G, Kaklamanis P, Lohmander S, Leeb B, Lequesne M, Mazieres B, Martin-Mola E, Pavelka K, Pendleton A, Punzi L, Serni U, Swoboda B, Verbruggen G, Zimmerman-Gorska I, Dougados M; Standing Committee for International Clinical Studies Including Therapeutic Trials ESCISIT. EULAR Recommendations 2003: an evidence based approach to the management of knee osteoarthritis: Report of a Task Force of the Standing Committee for International Clinical Studies Including Therapeutic Trials (ESCISIT). Ann Rheum Dis. 2003 Dec;62(12):1145-55. doi: 10.1136/ard.2003.011742. PMID 14644851
- [Background] National Board of Health, Denmark. Referenceprogram for knæartrose. Copenhagen: National Board of Health, Denmark; 2007. [22.02.2010] found at: http://www.sst.dk/publ/Publ2007/PLAN/SfR/Refprg_knaeartrose.pdf
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, part I: critical appraisal of existing treatment guidelines and systematic review of current research evidence. Osteoarthritis Cartilage. 2007 Sep;15(9):981-1000. doi: 10.1016/j.joca.2007.06.014. Epub 2007 Aug 27. PMID 17719803
- [Background] Walker-Bone K, Javaid K, Arden N, Cooper C. Regular review: medical management of osteoarthritis. BMJ. 2000 Oct 14;321(7266):936-40. doi: 10.1136/bmj.321.7266.936. No abstract available. PMID 11030685
- [Background] Hunter DJ, Felson DT. Osteoarthritis. BMJ. 2006 Mar 18;332(7542):639-42. doi: 10.1136/bmj.332.7542.639. No abstract available. PMID 16543327
- [Background] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen O, Rasmussen S. A Randomized, Controlled Trial of Total Knee Replacement. N Engl J Med. 2015 Oct 22;373(17):1597-606. doi: 10.1056/NEJMoa1505467. PMID 26488691
- [Derived] Skou ST, Roos E, Laursen M, Arendt-Nielsen L, Rasmussen S, Simonsen O, Ibsen R, Larsen AT, Kjellberg J. Cost-effectiveness of total knee replacement in addition to non-surgical treatment: a 2-year outcome from a randomised trial in secondary care in Denmark. BMJ Open. 2020 Jan 15;10(1):e033495. doi: 10.1136/bmjopen-2019-033495. PMID 31948990
- [Derived] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Rasmussen S, Simonsen O. Total knee replacement and non-surgical treatment of knee osteoarthritis: 2-year outcome from two parallel randomized controlled trials. Osteoarthritis Cartilage. 2018 Sep;26(9):1170-1180. doi: 10.1016/j.joca.2018.04.014. Epub 2018 May 1. PMID 29723634
- [Derived] Arendt-Nielsen L, Simonsen O, Laursen MB, Roos EM, Rathleff MS, Rasmussen S, Skou ST. Pain and sensitization after total knee replacement or nonsurgical treatment in patients with knee osteoarthritis: Identifying potential predictors of outcome at 12 months. Eur J Pain. 2018 Jul;22(6):1088-1102. doi: 10.1002/ejp.1193. Epub 2018 Feb 15. PMID 29369450
- [Derived] Skou ST, Roos EM, Simonsen O, Laursen MB, Rathleff MS, Arendt-Nielsen L, Rasmussen S. The effects of total knee replacement and non-surgical treatment on pain sensitization and clinical pain. Eur J Pain. 2016 Nov;20(10):1612-1621. doi: 10.1002/ejp.878. Epub 2016 Mar 31. PMID 27029553
- [Derived] Skou ST, Rasmussen S, Simonsen O, Roos EM. Knee Confidence as It Relates to Self-reported and Objective Correlates of Knee Osteoarthritis: A Cross-sectional Study of 220 Patients. J Orthop Sports Phys Ther. 2015 Oct;45(10):765-71. doi: 10.2519/jospt.2015.5864. Epub 2015 Aug 24. PMID 26304646
- [Derived] Skou ST, Roos EM, Laursen MB, Rathleff MS, Arendt-Nielsen L, Simonsen OH, Rasmussen S. Total knee replacement plus physical and medical therapy or treatment with physical and medical therapy alone: a randomised controlled trial in patients with knee osteoarthritis (the MEDIC-study). BMC Musculoskelet Disord. 2012 May 9;13:67. doi: 10.1186/1471-2474-13-67. PMID 22571284
- See also: Link to the published statistical analysis plan — http://vbn.aau.dk/da/publications/statistical-analysis-plan-sap-for-medic(120b4fb2-c21a-47f4-9255-ec9851a59f55).html

RESULTS

PARTICIPANT FLOW:
Groups:
- MEDIC: 60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Paracetamol: 1 g x 4/day
  Burana: 400 mg x 3/day
  Pantoprazol: 20mg x 1/day
  Dietary counseling: For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet.
  Patient education: The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA.
  Insoles: The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
- MEDIC + TKR: TKR: Surgical treatment with insertion of total knee replacement following standard procedures.
  Followed by:
  60min. of neuromuscular training two times a week for 3 months (12 weeks) using the neuromuscular training program called NEMEX-TJR.
  Paracetamol: 1 g x 4/day
  Burana: 400 mg x 3/day
  Pantoprazol: 20mg x 1/day
  Dietary counseling: For participants with a BMI equal to or >25. The dietitian initiates a 3-month intervention that provides instruction and guidance in relation to diet.
  Patient education: The aim is to strengthen the participant's involvement in the treatment, so the participant will be in a position to handle, master and act reasonable in relation to their knee OA.
  Insoles: The position of the knee is assessed using Single Leg Mini Squat. On the basis of this test it is decided which of two types of insoles (Formthotics System) the participant should have (neutral with a lateral wedge or neutral).
Period: Overall Study
Arm/Group | MEDIC | MEDIC + TKR
Started | 50 | 50
Completed | 49 | 46
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MEDIC | MEDIC + TKR | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.0 (8.7) | 65.8 (8.7) | 66.4 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 20 | 18 | 38
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.0 (5.8) | 32.3 (6.2) | 32.0 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in KOOS4 From Baseline (Knee Injury and Osteoarthritis Outcome Score)
Description: The average score for four of the five KOOS subscales, covering pain, symptoms, difficulties in functions of daily living, and quality of life (KOOS4), with scores ranging from 0 (worst) to 100 (best). Between group comparisons of treatment effect (change in KOOS4 from baseline to 1 year follow-up) will be dependent on data distribution. Between group comparisons of treatment effect (change in KOOS4 from baseline to 1 year follow-up) will be dependent on data distribution. We expect the change to be normally distributed and analysis will be made using a mixed model ANOVA with subject being a random factor and visit (baseline, 3, 6 and 12 months), treatment arm (TKA + MEDIC, MEDIC) and site (Frederikshavn, Farsoe) being fixed factors. Baseline KOOS4 will be a covariate. Furthermore interactions between the fixed factors will be included in the model. P-values and 95% CI will be presented to assess superiority.
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
units on a scale | 16.0 [10.1 to 21.9] | 32.5 [26.6 to 38.3]

2. Secondary Outcome: Change in EQ-5D From Baseline
Description: Between groups comparisons of the change from baseline to the 1 year follow-up in all secondary endpoint will be handled similar to the primary endpoint. See Statistical analysis plan for further description ("Links")
  Range of EQ-5D Descriptive Index is -0.59 to 1.00 (worst to best), while the EQ VAS goes from 0 to 100 (worst to best).
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
units on a scale
  Descriptive index | 0.115 [0.063 to 0.166] | 0.206 [0.141 to 0.270]
  Visual-analogue scale | 10.2 [4.6 to 15.7] | 15.0 [8.6 to 21.5]

3. Secondary Outcome: Change in Timed Up & Go (TUG) From Baseline
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: sec
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
sec | -1.2 [-1.8 to -0.6] | -2.4 [-3.1 to -1.6]

4. Secondary Outcome: Change in 20-meter Walk From Baseline
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: sec
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
sec | -1.0 [-1.5 to -0.4] | -2.9 [-3.8 to -1.9]

5. Secondary Outcome: Change in the Five Subscales of KOOS From Baseline
Description: All subscales going from 0 to 100 (worst to best)
Time Frame: Primary: 12months.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
units on a scale
  Pain | 17.2 [10.4 to 24.1] | 34.8 [28.1 to 41.5]
  Symptoms | 11.4 [4.4 to 18.4] | 26.4 [21.5 to 31.4]
  Activities of Daily Living | 17.6 [11.4 to 23.9] | 30.0 [22.7 to 37.2]
  Quality of Life | 17.8 [11.2 to 24.4] | 38.2 [30.6 to 45.8]
  Sports and recreation | 19.3 [10.8 to 27.7] | 34.5 [27.9 to 41.0]

6. Secondary Outcome: Weight Change in kg From Baseline
Description: Weight change in kg measured without shoes at the same time of day and on the same scale
Time Frame: Primary: 12months.
Population: Only patients with a BMI equal to or >25 were included in the analysis
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 43 | 39
kg | -2.6 [-3.9 to -1.4] | 0.1 [-1.5 to 1.7]

7. Secondary Outcome: Proportion of Users of Pain Medication
Description: With possible answers being yes and no
Time Frame: Baseline and 12months.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
proportion of participants
  Baseline | 0.58 [0.44 to 0.71] | 0.67 [0.53 to 0.79]
  12months | 0.41 [0.28 to 0.55] | 0.26 [0.15 to 0.41]

8. Secondary Outcome: Serious Adverse Events Related to the Index Knee
Description: Adverse events (AE) and seriously adverse events (SAE) will be registered in three ways and divided into index knee or sites other than index knee. The project physiotherapist will record any adverse events that the participant experiences or tells them about. For the participants allocated to, or crossing over to, TKA, a project worker will look through hospital records to register if any pre-defined perioperative and postoperative adverse events occurred. At all follow-ups, the assessor will use open-probe questioning to assess adverse events in all participants
Time Frame: Primary: 12months
Measure: Number; unit: Serious adverse events related to knee
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 50 | 50
Serious adverse events related to knee | 1 | 8

9. Other Pre Specified Outcome: Exploratory Outcomes
Description: 1. Pain intensities on a 100 mm VAS with terminal descriptors of 'no pain' and 'worst pain possible' in various situations.
  2. Number of sites with pain in the previous 24 hours shaded on a region-divided body chart
  3. Pain location and type assessed using the Knee Pain Map.
  4. Maximum isometric muscle strength (converted to Nm using the length of the lower leg) measured bilaterally in knee flexion and knee extension in a make test using a handheld dynamometer (Powertrack II TM Commander from JTech Medical Industries, Salt Lake City, Utah, USA)
  5. Pressure pain thresholds measured bilaterally using a handheld algometer (Algometer Type II, Somedic AB, Hoerby, Sweden)) at five sites at the knee and the m. tibialis anterior muscle.
  6. Self-efficacy in improving pain, function and QOL in various situations using a 100 mm VAS with terminal descriptors of 'very unsure' and 'very sure'.
  Further exploratory objectives may be added later on.
Time Frame: Baseline, 3months, 6months, 12months and 24 months.
Population: Will be reported in later publications, as it is exploratory outcomes
Arm/Group | MEDIC | MEDIC + TKR
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | MEDIC | MEDIC + TKR
Serious Adverse Events (participants affected / at risk) | 5/50 | 20/50
Other Adverse Events (participants affected / at risk) | 38/50 | 45/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=50) | MEDIC + TKR (N=50)
pain in the opposite knee leading to TKR (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoid tumor in the small intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
cerebral thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Stiffness requiring brisement forcé (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Deep infection in knee joint (Infections and infestations) | 0 (0) | 1 (1)
Deep venous thrombosis requiring anticoagulation (Vascular disorders) | 0 (0) | 3 (3)
femoral neck fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back pain leading to spinal fusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
abdominal pain with outpouching of the colon (Gastrointestinal disorders) | 0 (0) | 1 (1)
hiatal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
coronary thrombosis (Vascular disorders) | 1 (1) | 0 (0)
hospitalization due to suspicion of cerebral thrombosis caused by neurological symptoms in the legs (Vascular disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
hospitalization due to depression and anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
atrial fibrillation (Vascular disorders) | 0 (0) | 1 (1)
leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
hospitalization due to retinal detachment (Eye disorders) | 0 (0) | 1 (1)
trauma to the cranium from a fall leading to hospitalization (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
myelomatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MEDIC (N=50) | MEDIC + TKR (N=50)
Pain in index knee (Musculoskeletal and connective tissue disorders) | 21 (21) | 27 (27)
Swelling in index knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Instability of index knee (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Decreased range of motion of index knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6)
Joint distortion of index knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
sensation of the index knee locking up (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Calor and rubor around index knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
soft tissue calcification at index knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hospital care due to liquid oozing from the TKR scar (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
superficial infection of TKR knee (Infections and infestations) | 0 (0) | 1 (1)
bleeding from the TKR wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
numbness around the TKR scar (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
increased soreness around the TKR knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pruritus around the knee (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
serious illness in the family (Social circumstances) | 2 (2) | 1 (1)
lack of motivation/time (Social circumstances) | 2 (2) | 1 (1)
eye surgery (Eye disorders) | 1 (1) | 0 (0)
impaired balance (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
medication intake resulting in fatigue (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
advised by doctor to reduce the intensity of exercise due to hypertension (Social circumstances) | 1 (1) | 0 (0)
advised by doctor to exercise only once a week due to a lack of leukocytes (Social circumstances) | 1 (1) | 0 (0)
neuropathic wound on the foot (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
abscess in the gluteal region (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in the opposite knee (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
pain in the opposite knee with previous TKR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
pain in the hip (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
hand/finger surgery/fracture (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
painful pes planus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
sciatic nerve pain (Nervous system disorders) | 2 (2) | 0 (0)
low back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
rib, head and hip pain following two falls (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
short-lasting restless legs (Nervous system disorders) | 1 (1) | 2 (2)
paresthesia of the foot (Nervous system disorders) | 1 (1) | 0 (0)
shoulder surgery due to rupture of m. supraspinatus (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
lateral ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
ankle sprain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
pain in the hamstrings muscles (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Ankylosing Spondylitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
shoulder injury from a fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
muscle strain in the upper thigh (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
low haemoglobin percentage (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
abnormal swelling of the whole leg in the days after TKR surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
nausea (General disorders) | 0 (0) | 2 (2)
nerve pain (Nervous system disorders) | 0 (0) | 1 (1)
tranexamic acid given pre-surgery by mistake (unintended event) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
puncture of the synovial membrane during lateral release (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
mental unstability (Psychiatric disorders) | 0 (0) | 1 (1)
loss of consciousness leading to a fall (Vascular disorders) | 0 (0) | 1 (1)
lack of skin under the foot resulting in pain and limping (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
increased need of insulin (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Achilles tendinopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
iliotibial band syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
swelling of the foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
arm pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
muscle cramps (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
quadriceps strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
back and hip pain following a fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
pain in the hamstrings muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
short-lasting vertigo (Vascular disorders) | 0 (0) | 1 (1)
reduced walking distance (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No